CLINICAL TRIAL: NCT04196686
Title: Evaluating the Effectiveness of Immersive Technologies, Virtual Reality and Augmented Reality, to Increase Pain Threshold During Ice Immersion.
Brief Title: Ice Immersion Using Virtual Reality & Augmented Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 50951
Record Dates: First submitted 2019-11-19; First posted 2019-12-12 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-02

CONDITIONS: Pain, Neuropathic; Pain, Acute
Keywords: Virtual Reality; Augmented Reality; Ice Immersion
MeSH Terms: conditions — Neuralgia; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Ice bath Control then VR/AR (Experimental): Participants will be randomized with a 1:1 allocation to use their dominant or non-dominant hand with VR or control (no VR) for the cold pressor test and then crossed over. Participants will not be told of the specifics of the time limit, to avoid competitiveness and expectations and will be asked for pain scores every 30 seconds.
  Interventions: Device: VR/AR; Other: Ice Bath
- Ice bath with VR/AR then Control (Experimental): Participants will be randomized with a 1:1 allocation to use their dominant or non-dominant hand with VR or control (no VR) for the cold pressor test and then crossed over. Participants will not be told of the specifics of the time limit, to avoid competitiveness and expectations and will be asked for pain scores every 30 seconds.
  Interventions: Device: VR/AR; Other: Ice Bath

INTERVENTIONS:
Device: VR/AR — VR/AR headset with either passive or active content such as playing a game or watching a movie
Other: Ice Bath — Participants immerse hand in ice bath and starting again with their original assigned group and keep hand submerged as long as they can withstand the cold or until 4 minutes have elapsed, whichever comes first. Participants will not be told of the specifics of the time limit, to avoid competitiveness and expectations and will be asked for pain scores every 30 seconds.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of different technologies, Virtual Reality and Augmented Reality with modifications as passive content, active content, cognitive load modulation, and positive encouragement coaching to increase the pain threshold as assessed by immersing a hand in ice water.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* English speaking
* Hearing intact

Exclusion Criteria:

* Patients who do not consent
* Currently taking beta blockers or other chronotropic heart medication(s)
* Have a history of severe motion sickness
* Currently have nausea
* Currently experiencing seizures
* Are clinically unstable
* Have taken pain medications in the last 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 185 participants signed informed consent, 156 participants were allocated to a study arm
Groups:
- Ice Bath Control Then VR/AR: Participants placed their dominant or non-dominant hand in ice bath without the use of Virtual Reality (VR)/Augmented Reality (AR), then crossed to place their opposite hand in ice bath with the use of VR/AR
- Ice Bath With VR/AR Then Control: Participants placed their dominant or non-dominant hand in ice bath with the use of Virtual Reality (VR)/Augmented Reality (AR), then crossed to place their opposite hand in ice bath without the use of VR/AR
Period: First Treatment (4 Minutes)
Arm/Group | Ice Bath Control Then VR/AR | Ice Bath With VR/AR Then Control
Started | 78 | 78
Completed | 78 | 75
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3
Period: Second Treatment (4 Minutes)
Arm/Group | Ice Bath Control Then VR/AR | Ice Bath With VR/AR Then Control
Started | 78 | 75
Completed | 78 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis
Groups:
- All Participants: Participants placed their dominant or non-dominant hand in ice bath with or without the use of VR/AR, then crossed to place their opposite hand in ice bath using the opposite treatment or control
Arm/Group | All Participants
Number analyzed (Participants) | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.10 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 49
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 69
  More than one race | 12
  Unknown or Not Reported | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 153
First hand assignment [Count of Participants; unit: Participants]
  Dominant | 73
  Non-Dominant | 80
VR hand assignment [Count of Participants; unit: Participants]
  Dominant | 83
  Non-Dominant | 70

OUTCOME MEASURES:

1. Primary Outcome: VR Effect on Pain Tolerence
Description: Given that the cold pressor test produces an uncomfortable experience, we considered longer duration within the ice bath to represent increased pain tolerance. Measured in seconds (s).
Time Frame: Duration of ice bath (approximately 0 - 4 minutes)
Population: Participants who complete the respective interventions are included in the analysis.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Ice Bath Control: Participants placed their dominant or non-dominant hand in ice bath without the use of VR/AR
- Ice Bath With VR/AR: Participants placed their dominant or non-dominant hand in ice bath with the use of VR/AR
Arm/Group | Ice Bath Control | Ice Bath With VR/AR
Number analyzed (Participants) | 156 | 153
seconds | 135 (92) | 158 (89)
Statistical Analysis 1: Comparison: Ice Bath Control vs Ice Bath With VR/AR; Test type: Other; p < 0.001, Cox mixed effects model; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.25 to 0.51]

2. Secondary Outcome: VR's Effect on Perceived Pain Intensity
Description: During ice bath data collection participants will be asked to report pain on a numeric rating scale from 0-10, 0 being no pain and 10 being most excruciating pain imaginable every 30 seconds during ice bath
Time Frame: Duration of ice bath (approximately 0 - 4 minutes)
Population: Participants who complete the respective interventions are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ice Bath Control | Ice Bath With VR/AR
Number analyzed (Participants) | 156 | 153
score on a scale
  0 seconds | 2.1 (1.3) | 2.0 (1.3)
  30 seconds | 4.9 (2.1) | 4.4 (2.1)
  60 seconds | 6.0 (1.9) | 5.5 (2.0)
  90 seconds | 6.2 (2.0) | 5.9 (2.1)
  120 seconds | 6.0 (2.0) | 5.7 (2.0)
  150 seconds | 5.9 (2.0) | 5.5 (2.3)
  180 seconds | 5.6 (2.1) | 5.3 (2.4)
  210 seconds | 5.5 (2.3) | 5.1 (2.5)
  240 seconds | 5.2 (2.3) | 5.0 (2.6)
Statistical Analysis 1: Comparison: Ice Bath Control vs Ice Bath With VR/AR; Analysis was controlled for dominant hand treatment assignment, dominant hand order, and gender. Overall mean difference calculated from regression model; Test type: Other; p = 0.200, Linear mixed effects model; Mean Difference (Net) = 0.455, 95% CI 2-sided [0.32 to 0.59]

3. Secondary Outcome: Skin Conductance Response Density (SCRD)
Description: The effects of VR on modulating sympathetic response in the presence of painful stimuli, was assessed by analyzing SCRD per 30 second interval. We refer to each of these 30 second intervals as a separate epoch. Skin conductance is expected to increase with increasing sympathetic nervous system activity, as sympathetic activity increases sweat secretion to increase skin conductance.
Time Frame: Duration of ice bath (approximately 0 - 4 minutes)
Population: Participants who complete the respective interventions are included in the analysis.
Measure: Mean (Standard Deviation); unit: microsiemens
Arm/Group | Ice Bath Control | Ice Bath With VR/AR
Number analyzed (Participants) | 156 | 153
microsiemens | 0.10 (0.069) | 0.09 (0.061)
Statistical Analysis 1: Comparison: Ice Bath Control vs Ice Bath With VR/AR; The variables in the physiologic model were SCRD change over time and the SCRD change between groups, defined as those with and without VR; Test type: Other; p = 0.047, Linear mixed effects model; Mean Difference (Net) = 0.002, 95% CI 2-sided [0.00007 to 0.00368]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Ice Bath Control | Ice Bath With VR/AR
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/153
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/153
Other Adverse Events (participants affected / at risk) | 0/156 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT04196686/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT04196686/SAP_001.pdf